CLINICAL TRIAL: NCT05745077
Title: Using Data to Achieve Surgical Health Equity in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 852524
Record Dates: First submitted 2023-01-31; First posted 2023-02-27 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Gallbladder Disease
Keywords: Social Determinants of Health; Telemedicine; Elective Cholecystectomy; Emergency Cholecystectomy
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Consultation (Experimental): Patient will schedule a Telemedicine Consultation in place of traditional in-person visit.
  Interventions: Behavioral: Telemedicine Consultation
- Traditional In-Person Care (Active Comparator): Patient will schedule a traditional in-person visit as per usual care.
  Interventions: Behavioral: Traditional Care

INTERVENTIONS:
Behavioral: Telemedicine Consultation — Patients will be contacted by their surgeon over the phone to discuss surgical treatment.
  Arms: Telemedicine Consultation
Behavioral: Traditional Care — Patients will proceed with their surgical consultation as per standard practice.
  Arms: Traditional In-Person Care

SUMMARY:
The goal of this retrospective cohort and pragmatic pilot trial is to examine the social determinants of health in racial and ethnic minority patients from socially vulnerable backgrounds who have Gallbladder Disease (GBD). The main questions it aims to answer are:

1. What racial barriers in outcome exist for socially vulnerable patients with gallbladder disease?
2. How effective is telemedicine consultation in improving surgical outcomes for socially vulnerable patients with gallbladder disease?

Study participants will be asked to undergo telemedicine consultation in place of regular consultation with their doctor before undergoing treatment.

Researchers will compare the telemedicine consultation groups with traditional care patients to see if telemedicine consultation is effective at reducing surgical disparity outcomes.

DETAILED DESCRIPTION:
This study seeks to identify differences in the care paradigms to find and test solutions to racial disparities in emergent cholecystectomy, as well as develop and test a pilot study to compare the effectiveness of telemedicine consultation. To address surgical health equity in patients with gallbladder disease, this study aims to:

1. Examine racial disparities in outcomes of Primary Care Service Line (PCSL) patients with symptomatic GB disease with attention to conditional effects of social vulnerabilities (SV)
2. Compare the effectiveness study of telemedicine consultation for symptomatic GB disease in patients with social vulnerabilities

This study will be divided into two phases to address each aim. The first aim will be conducted as a retrospective cohort study and examine the outcomes of PCSL patients diagnosed with symptomatic GB disease between Jan. 1, 2020 and Sept. 30, 2022 using PennMedicine data to build regression models with interaction terms to examine racial disparities in surgical consultation and the conditional effects of SV factors on this relationship. The second aim will be performed as a pragmatic pilot trial of Penn PCSL patients with SV. For this aim, the investigators will pragmatically assign two groups to traditional care and telemedicine consultation and study the resultant outcomes from patients with diagnosed with symptomatic cholelithiasis or biliary colic as seen by a PCSL provider between April 1, and June 30, 2023. These results will provide data to develop evidence-based solutions to racial disparities within Penn Medicine and to serve as preliminary data for subsequent studies to promote health equity in patients with symptomatic GBD.

ELIGIBILITY:
Inclusion Criteria:

* Patients age > 18 in the Primary Care Service Line (PCSL) and Emergency Department (ED) discharges including referral to surgery
* Member of a racial or ethnic minority, not primary English speaking, from a low-income neighborhood, or underinsured
* With a new ICD-10 code for symptomatic cholelithiasis or biliary colic seen by a PCSL provider or discharge from an ED between February 1, and June 30, 2023

Exclusion Criteria:

* History of prior cholecystectomy
* Prisoner
* GB cancer
* Advanced cirrhosis
* Untreated coagulopathy
* No indication for surgery
* Unable/unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Cholecystectomy Surgical Outcome | 6 Months
  Compare rates of surgical consultation by consultation type.

SECONDARY OUTCOMES:
Time from Referral to Consultation | 6 Months
  Number of days between initial documentation of referral to surgery by provider and initial pre-operative consultation with surgeon by consultation type. Identified by EMR documentation and encounter visits.
Completion of Consultation | 6 Months
  Completion of initial pre-operative consultation visit with surgeon for patients referred to surgery. Identified by EMR documentation and encounter visits.
Effect of Consultation on Surgical Outcome. | 6 Months
  Operative treatment outcomes received by patients who received pre-operative consultation with the surgeon. Operative treatment will be determined using CPT and ICD-10-PCS codes for cholecystectomy as listed in HPM (CPT 47562, CPT 47563, CPT 47600, CPT 47605, CPT 56340, CPT 56341, ICD10 0FB40ZX, ICD10 OFB40ZZ, ICD10 OFT40ZZ).
Urgency of Operative Treatment | 6 Months
  Urgency for operative treatment for whether cholecystectomy was performed in the emergent or elective setting as determined by admission source for the associated operative encounter and CPT and ICD-10-PCS codes for cholecystectomy as listed in HPM (CPT 47562, CPT 47563, CPT 47600, CPT 47605, CPT 56340, CPT 56341, ICD10 0FB40ZX, ICD10 OFB40ZZ, ICD10 OFT40ZZ).
Cost | 6 Months
  Cost of care including preoperative consultation visit with the surgeon and cholecystectomy visit. Data will be obtained from Horizon Performance Manager.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Kelz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox, M.R., G.D. Eslick, and R. Padbury, The management of gallstone disease: a practical and evidence-based approach. 2018: Springer.
- [Background] Altieri MS, Yang J, Zhu C, Sbayi S, Spaniolas K, Talamini M, Pryor A. What happens to biliary colic patients in New York State? 10-year follow-up from emergency department visits. Surg Endosc. 2018 Apr;32(4):2058-2066. doi: 10.1007/s00464-017-5902-5. Epub 2017 Oct 23. PMID 29063306
- [Background] Prevention, C.f.D.C.a. Adult Obesity Facts. Division of Nutrition, Physical Activity, and Obesity, National Center for Chronic Disease Prevention and Health Promotion 2022 May 17, 2022 [cited 2022 September 19, 2022]; Available from: https://www.cdc.gov/obesity/data/adult.html#:~:text=Obesity%20affects%20some%20groups%20more%20than%20others&text=Non%2DHispanic%20Black%20adults%20(49.9,Hispanic%20Asian%20adults%20(16.1%25).%20Accessed%2009/18/2022.
- [Background] Overby DW, Apelgren KN, Richardson W, Fanelli R; Society of American Gastrointestinal and Endoscopic Surgeons. SAGES guidelines for the clinical application of laparoscopic biliary tract surgery. Surg Endosc. 2010 Oct;24(10):2368-86. doi: 10.1007/s00464-010-1268-7. Epub 2010 Aug 13. No abstract available. PMID 20706739
- [Background] Radunovic M, Lazovic R, Popovic N, Magdelinic M, Bulajic M, Radunovic L, Vukovic M, Radunovic M. Complications of Laparoscopic Cholecystectomy: Our Experience from a Retrospective Analysis. Open Access Maced J Med Sci. 2016 Dec 15;4(4):641-646. doi: 10.3889/oamjms.2016.128. Epub 2016 Nov 9. PMID 28028405
- [Background] Cheruvu CV, Eyre-Brook IA. Consequences of prolonged wait before gallbladder surgery. Ann R Coll Surg Engl. 2002 Jan;84(1):20-2. PMID 11892728
- [Background] Sobolev B, Mercer D, Brown P, FitzGerald M, Jalink D, Shaw R. Risk of emergency admission while awaiting elective cholecystectomy. CMAJ. 2003 Sep 30;169(7):662-5. PMID 14517123
- [Background] To KB, Cherry-Bukowiec JR, Englesbe MJ, Terjimanian MN, Shijie C, Campbell DA Jr, Napolitano LM. Emergent versus elective cholecystectomy: conversion rates and outcomes. Surg Infect (Larchmt). 2013 Dec;14(6):512-9. doi: 10.1089/sur.2012.160. Epub 2013 Nov 25. PMID 24274058
- [Background] Rutledge D, Jones D, Rege R. Consequences of delay in surgical treatment of biliary disease. Am J Surg. 2000 Dec;180(6):466-9. doi: 10.1016/s0002-9610(00)00520-1. PMID 11182399
- [Background] Munoz E, Tinker MA, Margolis I, Wise L. Surgonomics: the cost of cholecystectomy. Surgery. 1984 Oct;96(4):642-7. PMID 6435271
- [Background] Carmichael H, Moore A, Steward L, Velopulos CG. Using the Social Vulnerability Index to Examine Local Disparities in Emergent and Elective Cholecystectomy. J Surg Res. 2019 Nov;243:160-164. doi: 10.1016/j.jss.2019.05.022. Epub 2019 Jun 6. PMID 31177035
- [Background] Lin JA, Braun HJ, Schwab ME, Pierce L, Sosa JA, Wick EC. Pandemic Recovery: Persistent Disparities in Access to Elective Surgical Procedures. Ann Surg. 2023 Jan 1;277(1):57-65. doi: 10.1097/SLA.0000000000004848. Epub 2021 Mar 3. PMID 33914483
- [Background] Shenoy R, Kirkland P, Maggard-Gibbons M, Russell MM. Symptomatic Cholelithiasis: Do Minority Patients Experience Delays to Surgery? J Surg Res. 2022 Apr;272:88-95. doi: 10.1016/j.jss.2021.11.003. Epub 2021 Dec 22. PMID 34953371
- [Background] Janeway MG, Sanchez SE, Rosen AK, Patts G, Allee LC, Lasser KE, Dechert TA. Disparities in Utilization of Ambulatory Cholecystectomy: Results From Three States. J Surg Res. 2021 Oct;266:373-382. doi: 10.1016/j.jss.2021.03.052. Epub 2021 Jun 1. PMID 34087621
- [Background] Saluja S, Hochman M, Dokko R, Morrison JL, Valdez C, Baldwin S, Tandel MD, Cousineau M. Community-Based Health Care Navigation's Impact on Access to Primary Care for Low-Income Latinos. J Am Board Fam Med. 2022 Jan-Feb;35(1):44-54. doi: 10.3122/jabfm.2022.01.210253. PMID 35039411
- [Background] Han HR, Lee H, Kim MT, Kim KB. Tailored lay health worker intervention improves breast cancer screening outcomes in non-adherent Korean-American women. Health Educ Res. 2009 Apr;24(2):318-29. doi: 10.1093/her/cyn021. Epub 2008 May 7. PMID 18463411
- [Background] Chavarri-Guerra Y, Soto-Perez-de-Celis E, Ramos-Lopez W, San Miguel de Majors SL, Sanchez-Gonzalez J, Ahumada-Tamayo S, Viramontes-Aguilar L, Sanchez-Gutierrez O, Davila-Davila B, Rojo-Castillo P, Perez-Montessoro V, Bukowski A, Goss PE. Patient Navigation to Enhance Access to Care for Underserved Patients with a Suspicion or Diagnosis of Cancer. Oncologist. 2019 Sep;24(9):1195-1200. doi: 10.1634/theoncologist.2018-0133. Epub 2018 Nov 29. PMID 30498134
- [Background] Berkowitz RL, Phillip N, Berry L, Yen IH. Patient Experiences in a Linguistically Diverse Safety Net Primary Care Setting: Qualitative Study. J Particip Med. 2018 Jan 22;10(1):e4. doi: 10.2196/jopm.9229. PMID 33052110
- [Background] Gunter RL, Chouinard S, Fernandes-Taylor S, Wiseman JT, Clarkson S, Bennett K, Greenberg CC, Kent KC. Current Use of Telemedicine for Post-Discharge Surgical Care: A Systematic Review. J Am Coll Surg. 2016 May;222(5):915-27. doi: 10.1016/j.jamcollsurg.2016.01.062. Epub 2016 Feb 13. No abstract available. PMID 27016900
- [Background] Sathiyakumar V, Apfeld JC, Obremskey WT, Thakore RV, Sethi MK. Prospective randomized controlled trial using telemedicine for follow-ups in an orthopedic trauma population: a pilot study. J Orthop Trauma. 2015 Mar;29(3):e139-45. doi: 10.1097/BOT.0000000000000189. PMID 24983434
- [Background] Williams AM, Bhatti UF, Alam HB, Nikolian VC. The role of telemedicine in postoperative care. Mhealth. 2018 May 2;4:11. doi: 10.21037/mhealth.2018.04.03. eCollection 2018. PMID 29963556
- [Background] Hwa K, Wren SM. Telehealth follow-up in lieu of postoperative clinic visit for ambulatory surgery: results of a pilot program. JAMA Surg. 2013 Sep;148(9):823-7. doi: 10.1001/jamasurg.2013.2672. PMID 23842982
- [Background] Abbitt D, Choy K, Castle R, Carmichael H, Jones TS, Wikiel KJ, Barnett CC, Moore JT, Robinson TN, Jones EL. Telehealth follow-up after cholecystectomy is safe in veterans. Surg Endosc. 2023 Apr;37(4):3201-3207. doi: 10.1007/s00464-022-09501-6. Epub 2022 Aug 16. PMID 35974252
- [Background] Dekker PK, Bhardwaj P, Singh T, Bekeny JC, Kim KG, Steinberg JS, Evans KK, Song DH, Attinger CE, Fan KL. Telemedicine in the Wake of the COVID-19 Pandemic: Increasing Access to Surgical Care. Plast Reconstr Surg Glob Open. 2020 Dec 15;9(1):e3228. doi: 10.1097/GOX.0000000000003228. eCollection 2021 Jan. PMID 33564566
- [Background] Eruchalu CN, Bergmark RW, Smink DS, Tavakkoli A, Nguyen LL, Bates DW, Cooper Z, Ortega G. Demographic Disparity in Use of Telemedicine for Ambulatory General Surgical Consultation During the COVID-19 Pandemic: Analysis of the Initial Public Health Emergency and Second Phase Periods. J Am Coll Surg. 2022 Feb 1;234(2):191-202. doi: 10.1097/XCS.0000000000000030. PMID 35213441
- [Background] Maurer KR, Everhart JE, Ezzati TM, Johannes RS, Knowler WC, Larson DL, Sanders R, Shawker TH, Roth HP. Prevalence of gallstone disease in Hispanic populations in the United States. Gastroenterology. 1989 Feb;96(2 Pt 1):487-92. doi: 10.1016/0016-5085(89)91575-8. PMID 2642879
- [Background] Shaffer EA. Gallstone disease: Epidemiology of gallbladder stone disease. Best Pract Res Clin Gastroenterol. 2006;20(6):981-96. doi: 10.1016/j.bpg.2006.05.004. PMID 17127183
- [Background] Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care. 1998 Jan;36(1):8-27. doi: 10.1097/00005650-199801000-00004. PMID 9431328
- [Background] Kaufman EJ, Keele LJ, Wirtalla CJ, Rosen CB, Roberts SE, Mavroudis CL, Reilly PM, Holena DN, McHugh MD, Small D, Kelz RR. Operative and Nonoperative Outcomes of Emergency General Surgery Conditions: An Observational Study Using a Novel Instrumental Variable. Ann Surg. 2023 Jul 1;278(1):72-78. doi: 10.1097/SLA.0000000000005519. Epub 2022 Jul 4. PMID 35786573
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Schmidt M, Sondenaa K, Dumot JA, Rosenblatt S, Hausken T, Ramnefjell M, Njolstad G, Eide GE. Post-cholecystectomy symptoms were caused by persistence of a functional gastrointestinal disorder. World J Gastroenterol. 2012 Mar 28;18(12):1365-72. doi: 10.3748/wjg.v18.i12.1365. PMID 22493550
- [Background] Bell ML, Whitehead AL, Julious SA. Guidance for using pilot studies to inform the design of intervention trials with continuous outcomes. Clin Epidemiol. 2018 Jan 18;10:153-157. doi: 10.2147/CLEP.S146397. eCollection 2018. PMID 29403314
- [Derived] Bakillah E, Harbison S, Rosato FE, Altieri MS, Morris JB, Kaufman E, Schapira M, Peifer M, Kelz RR. Telemedicine and Access to Elective Cholecystectomy for Socially Vulnerable Adults: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2438137. doi: 10.1001/jamanetworkopen.2024.38137. PMID 39382898

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT05745077/Prot_SAP_000.pdf